CLINICAL TRIAL: NCT03186573
Title: Effect of Grape Juice Consumption on the Parameters of Oxidative Stress and Muscle Fatigue in Judo Athletes: A Randomized Clinical Trial
Brief Title: Effect of Grape Juice Consumption on the Parameters of Oxidative Stress and Muscle Fatigue in Judo Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Maria Júlia Vieira da Cunha Goulart, Nutricionist, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UFCSPAPortoAlegre
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-09

CONDITIONS: Oxidative Stress; Muscle Fatigue; Polyphenol; Free Radical Oxidation of Tissue
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The athletes will not receive any drink and will do the simulations of the fight.
- Intervention group (Active Comparator): (Intervention, grape juice) - athletes will receive 400 ml per day of grape juice (containing 66g of carbohydrates) for 14 days and will do the fight simulations.
  Interventions: Dietary Supplement: Grape juice
- Placebo Group (Placebo Comparator): (Placebo, grape-flavored maltodextrin carbohydrate) - athletes will receive400ml of drink daily with 66g of maltodextrin for 14 days and will do the fight simulations; The amount of maltodextrin is equal to the amount of carbohydrate present in grape juice.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Grape juice — 400ml diary of grape juice
  Arms: Intervention group
Dietary Supplement: Maltodextrin — 400ml diary of maltodextrin
  Arms: Placebo Group

SUMMARY:
This project aims to evaluate if after 14 days of grape juice ingestion there is improvement of the parameters of strength, fatigue and oxidative stress in judo fighters. The study will be a randomized, blind, crossover clinical trial of 20 Judo athletes. Judo wrestling simulations will be performed on 3 different days.

DETAILED DESCRIPTION:
Grape juice has a high concentration of phenolic compounds and is capable of modulating biochemical parameters and oxidative stress. By naturally containing carbohydrates grape juice can help acutely minimize fatigue during exercise as well as long-term oxidative stress parameters in athletes. This project aims to evaluate if after 14 days of grape juice ingestion there is improvement of the parameters of strength, fatigue and oxidative stress in judo fighters. The study will be a randomized, blind, crossover clinical trial of 20 Judo athletes. Judo wrestling simulations will be performed on 3 different days. Each exercise session will consist of four 7-minute bouts, with 14-minute rest between them. The athletes will perform a first fight simulation without ingestion of any beverage (control group 1), and then will be randomized to determine the order of participation in the groups: maltodextrin (group 2 placebo) and grape juice (intervention group 3). Analyzes of oxidative stress; Muscle strength and fatigue; Perceived effort rate; Lactate; Heart rate; Analysis of food consumption and body composition.Two-way ANOVA will be used to evaluate the relation of the intervention and physical exercise, besides parameters of strength and fatigue. The level of significance adopted will be 5% and for the analysis, the SPSS summer 23 statistical program will be used.

ELIGIBILITY:
Inclusion Criteria:

* Judo athletes, federated, who hold state, federal and international competitions of both sexes, aged between 15 and 24 years and any weight category of the sport, except free weight.

Exclusion Criteria:

* Recent injury (last 3 months) that prevents training or competition;
* Food restriction on grape juice;
* Being in the phase of fast weight loss in pre competition..

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Oxidative stress In Blood Collection | 15 days
  A disturbance in the prooxidant-antioxidant balance in favor of the former, leading to potential damage.

SECONDARY OUTCOMES:
Borg in scale. | 15 days
  Specific to muscle fatigue, a state arrived at through prolonged and strong contraction of a muscle. Studies in athletes during prolonged submaximal exercise have shown that muscle fatigue increases in almost direct proportion to the rate of muscle glycogen depletion. Muscle fatigue in short-term maximal exercise is associated with oxygen lack and an increased level of blood and muscle lactic acid, and an accompanying increase in hydrogen-ion concentration in the exercised muscle.

OTHER OUTCOMES:
Lactate in numbers | 15 days
  Specific to muscle fatigue, a state arrived at through prolonged and strong contraction of a muscle. Studies in athletes during prolonged submaximal exercise have shown that muscle fatigue increases in almost direct proportion to the rate of muscle glycogen depletion. Muscle fatigue in short-term maximal exercise is associated with oxygen lack and an increased level of blood and muscle lactic acid, and an accompanying increase in hydrogen-ion concentration in the exercised muscle.
Upper and lower limb strength in repetitions or numbers in meters | 15 days
  Specific to muscle fatigue, a state arrived at through prolonged and strong contraction of a muscle. Studies in athletes during prolonged submaximal exercise have shown that muscle fatigue increases in almost direct proportion to the rate of muscle glycogen depletion. Muscle fatigue in short-term maximal exercise is associated with oxygen lack and an increased level of blood and muscle lactic acid, and an accompanying increase in hydrogen-ion concentration in the exercised muscle.
Palmar grip strength - in strength and time | 15 days
  Specific to muscle fatigue, a state arrived at through prolonged and strong contraction of a muscle. Studies in athletes during prolonged submaximal exercise have shown that muscle fatigue increases in almost direct proportion to the rate of muscle glycogen depletion. Muscle fatigue in short-term maximal exercise is associated with oxygen lack and an increased level of blood and muscle lactic acid, and an accompanying increase in hydrogen-ion concentration in the exercised muscle.
muscle pain | 15 days
  Specific to muscle fatigue, a state arrived at through prolonged and strong contraction of a muscle. Studies in athletes during prolonged submaximal exercise have shown that muscle fatigue increases in almost direct proportion to the rate of muscle glycogen depletion. Muscle fatigue in short-term maximal exercise is associated with oxygen lack and an increased level of blood and muscle lactic acid, and an accompanying increase in hydrogen-ion concentration in the exercised muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Cláudia Dornelles Schneider, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Cláudia Dornelles Schneider, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided